CLINICAL TRIAL: NCT05595408
Title: Circulating and Urine Tumor DNA Dynamics Predict Minimal Residual Disease and Recurrence Risk in Locally Advanced Upper Tract Urothelial Carcinoma(CURATE-UTUC): A Multicenter Prospective Longitudinal Cohort Study
Brief Title: Circulating and Urine Tumor DNA Dynamics Predict Minimal Residual Disease and Recurrence Risk in Locally Advanced Upper Tract Urothelial Carcinoma
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CURATE-UTUC
Record Dates: First submitted 2022-10-22; First posted 2022-10-27 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Muscle Invasive Upper Tract Urothelial Carcinoma
Keywords: upper tract urothelial carcinoma; Minimal residual disease; Circulating tumor DNA; Urine tumor DNA; adjuvant chemotherapy; adjuvant immunotherapy
MeSH Terms: conditions — Neoplasm, Residual | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adjuvant chemotherapy group: muscle invasive upper tract urothelial carcinoma after radical nephroureterectomy receiving adjuvant chemotherapy
  Interventions: Drug: Adjuvant chemotherapy
- adjuvant immunotherapy group: muscle invasive upper tract urothelial carcinoma after radical nephroureterectomy receiving adjuvant immunotherapy
  Interventions: Drug: adjuvant immunotherapy

INTERVENTIONS:
Drug: Adjuvant chemotherapy — cisplatin/carboplatin-gemcitabine 4-6 cycles
  Groups: adjuvant chemotherapy group
Drug: adjuvant immunotherapy — immunotherapy for one year
  Groups: adjuvant immunotherapy group

SUMMARY:
In our study, the ultra-deep sequencing of circulating tumor DNA (ctDNA) and urine tumor DNA (utDNA) were performed to assess whether ctDNA and utDNA can be used as predictive biomarkers for the detection of minimal residual disease (MRD) and early diagnosis of UTUC recurrence, and explored the role of ctDNA and utDNA detection of MRD in the prediction of adjuvant therapy efficacy and prognostic evaluation.

DETAILED DESCRIPTION:
60% of Upper Urinary Tract Urothelial Carcinoma (UTUC) patients with muscle-invasive disease at diagnosis, which progresses rapidly, aggressively, and has a poor prognosis. Up to 30-40% of the patients may develop bladder recurrance after radical nephroureterectomy for primary upper tract urothelial carcinoma.

Minimal residual disease (MRD) refers to the small number of malignant cells that remain after curative treatments (curative intent surgical resection, radiotherapy, and/or chemotherapy). MRD is common in patients with blood cancer, and is known to be associated with recurrence and poor prognosis. Recent studies also reported that MRD-negative in postoperative solid tumors such as colorectal/colon cancer and muscle-invasive bladder cancer is associated with better survival outcomes. However, the clinical values of MRD monitoring for adjuvant therapy in postoperative UTUC remain inadequate.

A total of 84 patients with stage II-IV UTUC will be recruited in this clinical trial. The following plasma samples, urine samples and tumor tissues will be collected from each patient including T0 (preoperatively, 2[1-3] days before surgery), T1 (28±3 days postoperatively), T2 (within 7 days after cycle 2 adjuvant therapy), T3 (end-of-treatment), and quarterly/semi-annually during surveillance (T4-T6) until recurrence/24 months. In addition, demographic and tumor characteristics of the patients will be collected for subsequent analysis, including age, sex, tumor stage, pathological stage, disease couse time, etc. Tumor tissues and matched peripheral blood were collected before treatment and WES was used ctDNA detection techniques. For each patient, we selected up to 40 clonal somatic mutations for personalized, tumor informed ctDNA assay design.Statistical analyses will be performed to analyze the survival outcomes and to explore the clinical value of MRD monitoring for adjuvant therapy in postoperative UTUC.

ELIGIBILITY:
Inclusion Criteria:

* pathological comfirmed T2-4 or N+ and M0 upper tract urothelial carcinoma
* Male or female aged ≥18 years old who are willing to sign the informed consent form
* have no distant metastasis
* have an ECOG 0 to 2
* upper tract urothelial carcinoma patients received radical nephroureterectomy
* have no multiple primary carcinoma
* received adjuvant chemotherapy or immunotherapy after surgery within 12 weeks
* ≥2 postoperative liquid biopsy assessments (T1 and T2)

Exclusion Criteria:

* a prior history of bladder or synchronous bladder cancer
* Pregnant or lactating women, or patients who are fertile but do not take contraceptive measures;
* Severe infection;
* Severe heart disease;
* Uncontrollable neurological or mental disorders;
* Severe diabetes mellitus;
* Patients with severe autoimmune diseases.
* Neoadjuvant therapy exposure
* No bilateral UTUC
* Surveillance time < month
* <2 postoperative MRD surveillance assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pathological comfirmed T2-4 or N+ and M0 upper tract urothelial carcinoma patients who received adjuvant chemotherapy or immunotherapy after radical nephroureterectomy
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
extravesical recurrence free survival | 2 year
  The primary endpoint was extravesical recurrence-free survival (eRFS), defined as the time from radical nephroureterectomy (RNU) to the first occurrence of either locoregional recurrence (e.g., retroperitoneal lymph node, local soft tissue) or distant metastasis, as objectively confirmed by radiological imaging (CT or MRI) according to RECIST 1.1 criteria. Death from any cause without a prior documented extravesical recurrence was considered a competing risk event.

SECONDARY OUTCOMES:
Lead time of molecular recurrence detection | 2 year
  the interval from the first postoperative MRD-positive liquid biopsy to radiologic/cyotscopic
intravesical recurrence free survival | 2 year
  bladder or contralateral upper tract relapse confirmed by cystoscopy/ureteroscopy and biopsy
recurrence-free survival | 2 year
  Defined as the time from RNU to the first occurrence of any recurrence (including both extravesical and intravesical events).
Overall survival | 2 year
  efined as the time from RNU to death from any cause
Diagnostic performance of MRD assay | 2 year
  The sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of ctDNA (at T1, T2) for predicting extravesical recurrence, and of utDNA (at T2) for predicting intravesical recurrence, against the imaging and cystoscopic gold standards.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China